CLINICAL TRIAL: NCT06706583
Title: Clinical and Ecological Impact of a Primary Care Antimicrobial Stewardship Program Based on Telematic Educational Interviews. A Cluster Randomized Clinical Trial (TELÉMACO Trial)
Brief Title: Clinical and Ecological Impact of a Primary Care Antimicrobial Stewardship Program Based on Telematic Educational Interviews (TELÉMACO Trial)
Acronym: TELÉMACO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TELÉMACO
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Community Acquired Infections
Keywords: Antimicrobial Stewardship Program (ASP); Primary Care; Telemedicine; PIRASOA
MeSH Terms: conditions — Community-Acquired Infections

STUDY DESIGN:
Intervention Model Description: Cluster randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced education arm (Experimental): Telematic educational interviews are added to standard PIRASOA training
  Interventions: Behavioral: Telematic educational interviews + standard training
- Standard education arm (Active Comparator): Only standard PIRASOA training is provided
  Interventions: Behavioral: Standard training

INTERVENTIONS:
Behavioral: Telematic educational interviews + standard training — Physicians attending at healthcare centers in the experimental arm will receive periodic telematic educational interviews in which an Infectious Diseases consultant will provide practical training on the appropriate use of antibiotics through the review of one of the physician´s randomly chosen antibiotic prescription, according to a structured brief interview.
  In addition to this, each of these centres will continue carrying out the already established activities of the Regional ASP (PIRASOA).
  Arms: Enhanced education arm
Behavioral: Standard training — Primary Care Health Centers assigned to the control group will receive standard educational activities designated by the current Regional ASP (PIRASOA).
  Arms: Standard education arm

SUMMARY:
Brief Summary: Open-label, cluster randomized, multicenter clinical trial to evaluate the clinical and ecological impact of a Primary Care ASP based on telematic educational interviews.

DETAILED DESCRIPTION:
The objective of this project is to measure the effect of an Antimicrobial Stewardship Program (ASP) in Primary Care, based on an educational intervention.

This will consist of periodic structured telematic educational interviews between Infectious Diseases experts and Family Medicine and paediatrics specialists. In these interviews, the principles for the optimal use of antimicrobials will be addressed on real cases, analyzing together prescriptions randomly chosen from the Primary Care physician himself.

The repetition over time of key pedagogical messages for the optimisation of prescriptions is expected to improve the quality of antibiotic use, reduce the overall consumption, improve the use of microbiological tests, reduce the incidence of community infections caused by resistant microorganisms, and preserve patients' safety measured by the rate of admission for serious infections.

The results derived from these educational interventions, in the framework of a multimodal ASP, have been evaluated in hospital and Primary Care settings in quasi-experimental studies with a favourable outcome, but not in a clinical trial that specifically assesses the efficacy of educational interviews and avoids the bias of uncontrolled studies. To demonstrate this hypothesis, a cluster randomized trial has been designed, in wich all healthcare centers will be assigned either to a control group (the standard measures defined by the regional ASP PIRASOA will be maintained), and an experimental group (whose physicians will receive the educational intervention described).

ELIGIBILITY:
Inclusion criteria:

a) Primary Care centres within the reference area of the University Hospital Virgen del Rocío.

Exclusion criteria:

1. Emergency departments.
2. Odontology offices.
3. DDD per Health centre less than 5.78

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Total antimicrobial consumption | Monthly over a 36-month period
  Total antimicrobial antimicrobial will be measured using the recommended international standard, the Defined Daily Dose (DDD) per 1000 inhabitants per day.
  Predefined subgroup analyses will be conducted to assess the intervention's effect on the primary outcome based on: patient age, geneder, and socioeconomic level.

SECONDARY OUTCOMES:
Adequacy of antimicrobial prescriptions | Prevalence surveys will be performed at months +0, +7 and +15.
  The rate of appropriate antimicrobial prescriptions according to national reference guidelines will be assessed through three point prevalence surveys of randomly selected prescriptions.
Incidence density of hospitalizations due to infections | Monthly, over a 36-month period.
  The incidence density of hospitalizations due to infections (urinary, pneumonia and skin and soft tissue infections), and specifically due to Clostridiodes difficile infections per inhabitant.
Incidence density of resistant Enterobacterales in urine cultures | Monthly, over a 36-month period.
  Incidence density of resistant Enterobacterales in urine cultures per inhabitant sent from Primary Care centers from both arms.

CONTACTS AND LOCATIONS:
Overall Officials: José Miguel Cisneros Herreros, MD-PhD, Study Director — Hospitales Universitarios Virgen del Rocío
Locations (1):
- Hospital Universitario Virgen del Rocío, Seville, Spain

IPD SHARING:
Plan to Share IPD: Yes